CLINICAL TRIAL: NCT03441477
Title: Comparative Study of the NIDEK TONOREF III and the Haag-Streit Goldmann Manual Tonometer (Predicate) to Demonstrate Conformance to ANSI Z80.10-2014 Ophthalmic Instruments - Tonometers, to the FDA Guidance for Industry and FDA Staff, Tonometer-Premarket Notification [510(k)] Submissions, and to the Applicable Supplemental Information Sheet and Comparison of Pachymetry Values for NIDEK TONOREF III With the NIDEK CEM-530 (Predicate)
Brief Title: Comparative Study of the NIDEK TONOREF III and the Haag-Streit Goldmann Manual Tonometer and Comparison of Pachymetry Values for NIDEK TONOREF III With the NIDEK CEM-530
Status: Completed | Type: Interventional
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIDEK-TONOREF-US-0001
Record Dates: First submitted 2018-01-17; First posted 2018-02-22 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2022-01

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Adults 18 years old or older (Experimental): Nidek Tonoref III
  Interventions: Device: Nidek Tonoref III; Device: Haag-Streit Goldmann Manual Tonometer; Device: NIDEK CEM-530

INTERVENTIONS:
Device: Nidek Tonoref III — The auto ref/kerato/tono/pachymeter TONOREF III is a medical device which measures objective refractive errors, corneal curvature radius, intraocular pressure and corneal thickness of the patient's eye.
Device: Haag-Streit Goldmann Manual Tonometer — Haag-Streit Goldmann Manual Tonometer measures intraocular pressure to aid in the screening and diagnosis of glaucoma
Device: NIDEK CEM-530 — Nidek CEM-530 is a non-contact ophthalmic microscope, optical pachymeter, and camera used for examination of the corneal endothelium and for measurement of the thickness of the cornea.

SUMMARY:
The primary objective of this clinical study is to prove that tonometry values for NIDEK TONOREF III are comparable to the predicate device and to prove that the pachymeter function of NIDEK TONOREF III is equivalent to the predicate device. The secondary objective is to demonstrate that the test device is as safe as the predicate devices.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years of age of either sex and any race or ethnicity;
2. be willing and able to provide written informed consent prior to any study procedures being performed;
3. be willing and able to follow all instructions and attend all study visits;

Exclusion Criteria:

1. have only one functional eye;
2. have poor or eccentric fixation in either eye;
3. have corneal scarring or have had corneal surgery, including corneal laser surgery in either eye;
4. have microphthalmos in either eye;
5. have buphthalmos in either eye;
6. be a contact lens wearer, meaning having worn soft contact lenses within the past 3 months and/or rigid permeable gas lenses within the past 6 months;
7. have dry eyes, meaning having been diagnosed by a physician with dry eyes and currently using a prescribed medication or daily use of artificial tears;
8. be a lid squeezer - blepharospasm;
9. have nystagmus in either eye;
10. have keratoconus in either eye;
11. have any other corneal or conjunctival pathology or infection in either eye;
12. have a condition or a situation, which in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NIDEK TONOREF III Comparison: Adults, 18 years old or older, were enrolled in this study. Participants were measured by the NIDEK TONOREF III and the Haag-Streit GAT and the NIDEK CEM-530, or the NIDEK TONOREF III and the NIDEK CEM-530.
Period: Overall Study
Arm/Group | NIDEK TONOREF III Comparison
Started | 225
Completed | 224
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: A total of 225 subjects were enrolled in the study and comprised the safety population; 224 subjects completed the study. One subject was discontinued due to a protocol violation. 223 subjects were included in the CCT Efficacy Subpopulation. One subject was excluded from the CCT Efficacy Subpopulation due to unevaluable results.
Arm/Group | NIDEK TONOREF III Comparison
Number analyzed (Participants) | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 210
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 46
  White | 168
  More than one race | 1
  Unknown or Not Reported | 0
Iris Color [Count of Participants; unit: Participants]
  Black | 8
  Blue | 49
  Brown | 126
  Hazel | 28
  Green | 10
  Grey | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Agreement of Intraocular Pressure
Description: Agreement of the measured IOP between the test device and the predicate device for the tonometer function of NIDEK TONOREF III.
  The mean difference and the standard deviation between these two devices are shown in the outcome measures table.
Time Frame: 1 day
Population: Data of subjects with 500-600µm CCT and ≤3D Astigmatism.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- NIDEK TONOREF III Comparison: IOP value were compared between NIDEK TONOREF III and Haag-Streit GAT
Arm/Group | NIDEK TONOREF III Comparison
Number analyzed (Participants) | 120
mmHg | 0.3 (3.45)

2. Primary Outcome: Agreement of Corneal Thickness
Description: Agreement of the measured corneal thickness between the test device and the predicate device for the pachymeter function of the NIDEK TONOREF III.
  The mean difference and the standard deviation between these two devices are shown in the outcome measure table.
Time Frame: 1 day
Population: Subjects with 300-800 μm CCT (Predicate)
Measure: Mean (Standard Deviation); unit: μm
Groups:
- NIDEK TONOREFIII Comparison: CCT were compared between NIDEK TONOREF III and NIDEK CEM-530.
Arm/Group | NIDEK TONOREFIII Comparison
Number analyzed (Participants) | 223
μm | -7.1 (8.31)

3. Secondary Outcome: Number of Occurrences of Adverse Events
Description: Any sight threatening adverse event associated with the test and predicate devices.
Time Frame: 1day
Population: Adverse Events were monitored irrespective of specific device and therefore cannot be separated.
Measure: Count of Participants; unit: Participants
Groups:
- NIDEK TONOREF III Comparison: Adverse Events were monitored irrespective of specific device and therefore cannot be separated.
Arm/Group | NIDEK TONOREF III Comparison
Number analyzed (Participants) | 225
Participants | 1

ADVERSE EVENTS:
Time Frame: 1day
Arm/Group | NIDEK TONOREF III Comparison
All-Cause Mortality (participants affected / at risk) | 0/225
Serious Adverse Events (participants affected / at risk) | 0/225
Other Adverse Events (participants affected / at risk) | 1/225
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIDEK TONOREF III Comparison (N=225)
Punctate epithelial erosions (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03441477/Prot_SAP_001.pdf